CLINICAL TRIAL: NCT04314908
Title: The Clinical Comparative Evaluation of Sonic Activation Assisted Irrigation and Apical Enlargement on Postoperative Endodontic Pain In Retreatment: A Prospective Randomized Clinical Trial
Brief Title: "Effect of Sonic Activation Assisted Irrigation and Apical Enlargement on Postoperative Endodontic Pain"
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 224
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2020-05-01 (Actual); Status verified 2020-03

CONDITIONS: Postoperative Pain; Endodontically Treated Teeth
Keywords: Endodontics; Postoperative Pain; Visual Analogue Pain Scale
MeSH Terms: conditions — Pain, Postoperative; Tooth, Nonvital

STUDY DESIGN:
Intervention Model Description: Parallel Assignment The patients were assigned to 4 medication groups randomly with an equal allocation rate between groups.The patients in the groups had same characteristics.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant and Outcomes Assessor) The patients and outcome assessor were unaware as to which study group they had been allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Apical enlargement (Experimental): Routine retreatment procedure will be performed at working length according to the apex locator at point "0".
  Interventions: Procedure: Apical enlargement
- Apical enlargement + Sonic Activation Assisted Irrigation (Experimental): Routine retreatment procedure will be performed at working length according to the apex locator at point "0" and sonic activation assisted irrigation will be applied.
  Interventions: Procedure: Apical enlargement + Sonic Activation Assisted Irrigation
- Non Apical enlargement (Experimental): Routine retreatment procedure will be performed at working length according to the apex locator at 1mm shorter than "0" point.
  Interventions: Procedure: Non Apical enlargement
- Non Apical enlargement + Sonic Activation Assisted Irrigation (Experimental): Routine retreatment procedure will be performed at working length according to the apex locator at 1mm shorter than "0" point and sonic activation assisted irrigation will be applied.
  Interventions: Procedure: Non Apical enlargement + Sonic Activation Assisted Irrigation

INTERVENTIONS:
Procedure: Apical enlargement — The teeth in this group will be treated according to the guidelines for retreatment in single-session. The filling will remove and cavity will be opened. The working length will be measured using apex locator and the "0" point will be based on. After standard irrigation protocol, root canals will be obturated with gutta percha and root canal sealer. Coronal restoration will complete using composite and/or fully crown if necessary.
  Arms: Apical enlargement
Procedure: Apical enlargement + Sonic Activation Assisted Irrigation — The teeth in this group will be treated according to the guidelines for retreatment in single-session. The filling will remove and cavity will open. The working length will be measured using apex locator and the "0" point will be based on. After standard irrigation protocol, sonic activation assisted irrigation will be applied to the root canals. Then the teeth were obturated with gutta percha and root canal sealer. Coronal restoration will complete using composite and/or fully crown if necessary.
  Arms: Apical enlargement + Sonic Activation Assisted Irrigation
Procedure: Non Apical enlargement — The teeth in this group will be treated according to the guidelines for retreatment in single-session. The filling will remove and cavity will open. The working length will be measured using apex locator and 1 mm shorter than the "0" point will be based on. After standard irrigation protocol, root canals will be obturated with gutta percha and root canal sealer. Coronal restoration will complete using composite and/or fully crown if necessary.
  Arms: Non Apical enlargement
Procedure: Non Apical enlargement + Sonic Activation Assisted Irrigation — The teeth in this group will be treated according to the guidelines for retreatment in single-session. The filling will remove and cavity will open. The working length will be measured using apex locator and 1 mm shorter than the "0" point will be based on. After standard irrigation protocol, sonic activation assisted irrigation will be applied to the root canals. Then the teeth were obturated with gutta percha and root canal sealer. Coronal restoration will complete using composite and/or fully crown if necessary.
  Arms: Non Apical enlargement + Sonic Activation Assisted Irrigation

SUMMARY:
The purpose of this randomized clinical trial is to evaluate the incidence of postoperative pain after retreatment after apical enlargement and sonic activation assisted irrigation. The presence of postoperative pain will assess after retreatment cases at 12, 24, 48, 72 hrs and 1 week.

DETAILED DESCRIPTION:
The aim of this clinical study is to evaluate the intensity and duration of postoperative pain after apical enlargement and sonic activation assisted irrigation procedures. Patients who have asymptomatic teeth required retreatment will include in this study and retreatment procedure will be applied to these teeth. One hundreds twenty asymptomatic teeth required retreatment will randomly participate into 4 treatment groups in terms of apical enlargement and sonic activation assisted irrigation procedure applied. The presence of postoperative pain will assess after 12, 24, 48, 72 hrs and 1 week. Postoperative pain will be recorded by each patient by using visual analogue pain scale. Before the treatments, the nature of the study, complications and associated risks will be totally explained and written informed consent will be obtained from all study participants. The local anesthetic will be applied before the treatment start. The routine retreatment procedure will be applied. Different final irrigation solutions will be applied in accordance to the manufacturers' instructions. At the end of treatment, each patient will be given an evaluation sheet, explained the treatment procedure and using of visual analogue pain scales, and informed to be returned during the following one week. After one week the teeth will be examined according to for pain intensity, percussion & palpation sensitivity, swelling, analgesic intake and clinical status.

ELIGIBILITY:
Inclusion Criteria:

-Patients who were healthy volunteers and who have failed teeth required retreatment with periapical index score 3-5 score requiring root canal treatment for first time.

Patients who were not included the study who;

* were pregnant or breast feeding during the duration of the study,
* have systemic disease, have any pain and/or any facial swelling, abscess,
* were immunocompromised,
* were under 18 yrs. and over 65 yrs. age,
* were taking antibiotics or corticosteroids within previous three days,
* have multiple teeth that required root canal treatment at the same time period; for eliminating pain referral,
* have root canals that could not be well-treated with orthograde retreatment.

Exclusion Criteria:

-The patients who forgot to fill out the form and took antibiotics and/or analgesics right after the first appointment of the therapy were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-10 (Estimated); Primary Completion 2020-10-10 (Estimated); Study Completion 2021-12-10 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Postoperative Pain after Root Cana Treatment at 1 week: VAS | Baseline, 12, 24, 48, 72 hours and 1 week.
  The primary outcome measure of the study is to assess if sonic activation assisted irrigation and apical enlargement procedures influence the occurrence of postoperative pain.Postoperative pain was assessed using a well defined Heft-Parker visual analogue scale (VAS) scale. Each patient recorded the pain level on a 100-mm VAS scale experimental basis for revising the graphic rating scale for pain in well-defined categories at 5 time intervals as 12, 24, 48, 72 hours and 1 week after treatment. The VAS scale was divided into 4 categories: No pain or faint pain corresponded to 0 mm. Mild pain was defined as greater than 0 mm and less than or equal to 25 mm. Mild pain included the descriptors of weak and mild pain. Moderate pain was defined as greater than 50 mm and less than 75 mm. Intense pain was defined as equal to or greater than 75 mm. Intense pain included the descriptors of strong, severe, and maximum possible.

CONTACTS AND LOCATIONS:
Overall Officials: Keziban Olcay, DDS, Phd, Principal Investigator — Medipol University